CLINICAL TRIAL: NCT04310085
Title: A Single Centre, Open Label, Pilot Phase Ib Study to Investigate Blood Stage Malaria Infection After Direct Venous Inoculation of Cryopreserved P. Falciparum (NF54 Strain) Sporozoites (PfSPZ-DVI) in Malaria naïve Healthy Adult Volunteers
Brief Title: Study in Blood Stage Malaria Infection After DVI of Cryopreserved P. Falciparum (NF54 Strain) Sporozoites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other); Institute of Tropical Medicine, Belgium (Other); Swiss BioQuant (Industry); PrimeVigilance Ltd., UK (Industry); Sanaria Inc. (Industry); Iqvia Pty Ltd (Industry); FGK Representative Service B.V., The Netherlands (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PfSPZ-DVI Blood Stage_19_01; 2019-004317-14 (EudraCT Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Malaria,Falciparum; Parasitemia; Protozoan Infections; Parasitic Disease
Keywords: Malaria; PfSPZ Challenge
MeSH Terms: conditions — Malaria, Falciparum; Parasitemia; Protozoan Infections; Parasitic Diseases; Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: All subjects will receive the PfSPZ Challenge product. In cohort 1 parasitaemia will be allowed to develop until a threshold of 5000 parasites/mL blood or a malaria clinical score ≥6 is reached. In cohort 2 the threshold is 10 000/mL or a malaria clinical score of ≥6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PfSPZ-DVI challenge and artemether lumefantrine (Experimental): 16 healthy, malaria-naïve males and females, aged 18-55 years, were enrolled in 2 cohorts (8 participants/cohort; a participant may be enrolled in one cohort only). There were two target levels of parasitaemia previously achieved in healthy participants in malaria VIS at other study sites, i.e., 5000 parasites/mL blood in Cohort 1 and 10000 parasites/mL blood in Cohort 2. (Based on observed levels of parasitaemia in Cohort 1, the target threshold for treatment in Cohort 2 was maintained at 5,000 p/mL).
  qPCR was performed, malaria clinical score assessed twice daily and participants were administered registered antimalarial therapy, i.e., Riamet®, when the following criteria were met:
  1. Cohort 1: ≥5000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
  2. Cohort 2: ≥10000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
  Interventions: Drug: Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet; Biological: PfSPZ-DVI Challenge

INTERVENTIONS:
Drug: Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet — artemether-lumefantrine 6 x of 4 tablets at approximately 0, 8, 24, 36, 48 and 60 h
  Other Names: Riamet
Biological: PfSPZ-DVI Challenge — 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)

SUMMARY:
This is a single-centre, open-label, Phase Ib study designed to assess if intravenous injection of approximately 3200 P. falciparum (NF54 strain) sporozoites can be safely administered to achieve blood-stage parasitaemia with a kinetics/PCR profile that will allow for the future characterisation of antimalarial blood-stage activity of new chemical entities in a relatively small number of participants during early drug development.

Healthy, malaria-naïve adults, aged 18-55 years, will be enrolled in a maximum of 2 cohorts. Enrolment into the cohorts will proceed sequentially, with two target levels of parasitaemia, i.e., 5000 parasites/mL blood in Cohort 1 and 10000 parasites/mL blood in Cohort 2.

(Based on observed levels of parasitaemia in Cohort 1, the target threshold for treatment in Cohort 2 was maintained at 5,000 p/mL (vs 10,000 p/mL in the protocol)).

The 3-day antimalarial therapy regimen will be further administered and monitored until parasite clearance. Safety and tolerability will be monitored during the whole study duration.

DETAILED DESCRIPTION:
Up to 16 healthy, malaria-naïve males and females, aged 18-55 years, will be enrolled in a maximum of 2 cohorts (up to 8 participants per cohort; a participant may be enrolled in one cohort only). Enrolment into the cohorts will proceed sequentially, with two target levels of parasitaemia previously achieved in healthy participants enrolled in malaria Volunteer Infection Studies (VIS) at other study sites, i.e., 5000 parasites/mL blood in Cohort 1 and 10000 parasites/mL blood in Cohort 2. (Based on observed levels of parasitaemia in Cohort 1, the target threshold for treatment in Cohort 2 was maintained at 5,000 p/mL (vs 10,000 p/mL in the protocol)).

Each participant will be admitted to the clinical unit in the morning of Day -1 and inoculated with approximately 3200 P. falciparum sporozoites (NF54 strain) by DVI on Day 1. Participants will be discharged 2 h post inoculation on Day 1 and will be monitored daily via phone call from Day 2 until Day 6 to solicit any AEs. Participants will come to the clinical unit daily from Day 7 until Day 9 and together with the malaria clinical score (see Attachment 1), the presence of parasites will be assessed once daily by a specific qPCR targeting the varATS (the acidic terminal segment in Plasmodium falciparum var genes) multigenic family; this to accurately describe parasite growth even in case PCR positivity, i.e., a qPCR outcome ≥250 parasites per mL blood, is confirmed this early (very low probability and with low densities). Participants will be confined to the clinical unit from Day 10 in the morning. qPCR will be performed and malaria clinical score assessed twice daily and participants will be administered registered antimalarial therapy, i.e., Riamet®, when the following criteria are met:

1. Cohort 1: ≥5000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
2. Cohort 2: ≥10000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.

The registered 3-day antimalarial therapy regimen will be further administered and monitored. qPCR assessments of parasitaemia will be carried out at multiple time points (2, 6, 8, 12, 16, 24, 36, 48 and 72 h) following initiation of Riamet® and malaria clinical score will be assessed twice daily during confinement in the clinical unit. Safety and tolerability will be monitored during the whole study duration, specific assessments will be done at periodic pre-specified time points from Day 10 and for at least 72 h after initiating antimalarial therapy, i.e., during confinement in the clinical unit (see below).

Of note, all participants must consent to receiving antimalarial therapy, i.e., the registered 3-day Riamet® regimen approved for treatment of uncomplicated malaria. Even in the case of withdrawal from the study, all participants administered the PfSPZ-DVI Challenge are to receive antimalarial therapy as soon as possible, and to have all appropriate visits and assessments as required. If an intolerance or contraindication to Riamet® develops, Malarone® will be administered.

Upon parasite clearance (defined as a qPCR value of 0 parasites per mL blood after initiating antimalarial therapy) and at least 72 h after initiating antimalarial therapy (estimated to occur on or before Day 19 and on or before Day 22 for Cohort 1 and Cohort 2, respectively), and if clinically well, participants will be discharged from the clinical unit and will be followed up for safety assessments, clinical evaluation and malaria qPCR in the clinical unit at the EOS visit on Day 28. All participants who received antimalarial therapy will be asked non-leading questions to determine the occurrence of any AEs throughout the study and at the EOS visit. All participants inoculated with PfSPZ-DVI Challenge will commence antimalarial therapy no later than Day 24 for both cohorts, regardless if they reach pre-defined cohort-specific PCR parasitaemia/malaria clinical score thresholds (i.e., 5000 parasites/mL blood for Cohort 1 and 10000 parasites/mL blood for Cohort 2 and/or a malaria clinical score ≥6 for Cohorts 1 and 2). Participants who start antimalarial therapy on Day 24 will only be discharged from confinement at the end of the EOS visit on Day 28. Antimalarial therapy may be initiated whenever deemed necessary by the Investigators, e.g., if there is a concern regarding the safety of a study participant. Therapy may be amended according to the treating physician if the participant does not respond to treatment or the condition worsens.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent Form signed voluntarily before any study-related procedure is performed, indicating that the participant understands the purpose of and procedures required for the study and is willing to participate in the study, including administration of registered antimalarial therapy;
2. Male or female, between 18 and 55 years old (extremes included) at screening;
3. Body weight of at least 50 kg and a body mass index (BMI) of 19.0 to 30.0 kg/m2 (extremes included);
4. Good general health without clinically relevant medical illness, physical exam findings including vital signs, and laboratory abnormalities (e.g., without liver transaminases >1x ULN and according to the clinically acceptable ranges for study inclusion laboratory tests in Attachment 4) as determined by the Investigator;
5. Willing to adhere to the prohibitions and restrictions specified in this protocol (see Section 4.3), including willingness to stay confined to the inpatient unit for the required duration and willingness to avoid travelling outside of Benelux during the study period;
6. Female participants should fulfil one of the following criteria:

   1. At least 1 year postmenopausal (amenorrhea >12 months and follicle-stimulating hormone [FSH] >30 mIU/mL) prior to screening;
   2. Surgically sterile (bilateral oophorectomy, hysterectomy or bilateral salpingectomy);
   3. Will use contraceptives as outlined in inclusion criterion 7;
7. Female participants of childbearing potential (excluding females with female partners) must agree to the use of a highly effective method of birth control from the screening visit until 40 days after the EOS visit at Day 28 (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose of Riamet®); Note: Highly effective birth control methods include: combined (oestrogen- and progestogen-containing) oral/intravaginal/transdermal hormonal contraception associated with inhibition of ovulation, progestogen-only oral/injectable/implantable hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence from heterosexual intercourse.
8. Female participant has a negative pregnancy test at screening and upon admission in the clinical unit; Note: Pregnancy testing will consist of serum β-human chorionic gonadotropin (β-HCG) tests at screening and at the EOS visit and a urine β-HCG tests on Day -1, in all women.
9. Different ways of being reachable 24/7 (e.g., by mobile phone, regular phone or electronic mail) during the whole study period.

Exclusion Criteria:

* 1. Nursing (lactating) women; 2. Participation in any other clinical drug or vaccine study within 30 days (or 5 half-lives for drugs) preceding the day of PfSPZ-DVI Challenge (whichever is longer), or plans to participate in other investigational drug or vaccine research during the study period; 3. Participants who took standard vaccinations within 3 months before the start of the study or are planning to take standard vaccinations during the study period up to 8 weeks after PfSPZ-DVI Challenge; 4. Blood product donation to any blood bank during the 8 weeks (whole blood) or 4 weeks (plasma and platelets) prior to admission in the clinical unit on Day -1; 5. Mean ECG outside normal range and deemed clinically relevant by the Investigator. Examples of clinically significant ECG abnormalities for this study include:
* PR-interval >220 ms;
* QRS-complex >120 ms;
* Absolute QT greater than >500 ms;
* QT interval corrected according to Bazett's formula (QTcB) or QTcF >450 ms for male participants, >470 ms for female participants;
* Pathologic Q wave;
* Significant ST-T wave changes;
* Left or right ventricular hypertrophy;
* Non-sinus rhythm except isolated premature atrial contractions and ventricular extrasystole <2 per 10 s ECG lead;
* Incomplete left bundle branch block, or complete or intermittent right or left bundle branch block;
* Second or third degree A-V heart block. 6. Seropositive human immunodeficiency virus (HIV), hepatitis A immunoglobulinM (IgM) antibody, hepatitis B virus (HBV) (hepatitis B surface antigen [HBsAg]), hepatitis C virus (HCV) (antibody), hepatitis D antibody, hepatitis E IgM antibody, cytomegalovirus (CMV) IgM antibody or Epstein Barr Virus (EBV) IgM antibody; 7. Previous or current diagnosis of hepatitis including but not limited to viral hepatitis, auto-immune hepatitis, non-alcoholic steatohepatitis (NASH), alpha-1-antitrypsin deficiency, alcoholic liver disease, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), hemochromatosis, Wilson disease or suspected hepatocellular carcinoma (HCC).

  8. History or presence of diagnosed food or known drug allergies (including but not limited to allergy to any of the antimalarial medications to be used in the study, see Section 5.1), or history of anaphylaxis or other severe allergic reactions; Note: Participants with seasonal allergies/hay fever, house dust mite or allergy to animals that are untreated and asymptomatic at the time of dosing can be enrolled in the study.

  9. History of convulsion or severe head trauma, excluding fever convulsion under 5 years of age; Note: A medical history of a single febrile convulsion during childhood is not an exclusion criterion.

  10. History of serious psychiatric condition that may affect participation in the study or preclude compliance with the protocol, including but not limited to past or present psychoses, disorders requiring lithium, a history of attempted or planned suicide, more than one previous episode of major depression, any previous single episode of major depression lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening; Note: The Beck Depression Inventory (Attachment 2) will be used as an objective tool for the assessment of depression at screening. In addition to the conditions listed above, participants with a score of 20 or more on the Beck Depression Inventory and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. Participants with a Beck score of 17 to 19 may be enrolled at the discretion of the Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the volunteer or to the execution of the study and interpretation of the data gathered.

  11. A medical, occupational or family problem as a result of alcohol or illicit drug abuse during the past 12 months or current alcohol or illicit drug abuse or addiction (positive alcohol breath test or positive drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine or opiates at screening or upon check-in at the clinical unit); Note: Excessive use of alcohol is defined as an intake of >21 units per week for males and >14 units per week for females where one alcohol unit is defined as 10 mL or 8 g of pure alcohol. A single unit is equal to one 25-mL (single) measure of whisky (alcohol by volume [ABV] 40%), or a third of a pint of beer (190 mL; ABV 5-6%) or half a standard (175 mL) glass of wine (ABV 12%).

  12. Participants are non-smokers or ex-smokers for more than 90 days prior to screening, or smoke no more than 5 cigarettes per day. If users of nicotine products (i.e., spray, patch, e-cigarette, etc.), they should use the equivalent of no more than 5 cigarettes per day. Participants must agree to abstain from smoking while in the unit; 13. Use of any prescription drugs, herbal supplements (e.g., St John's Wort) or over-the-counter medication within 7 days or 5 half-lives (whichever is longer) prior to the PfSPZ-DVI Challenge, or an anticipated requirement for the use of these during the course of the study (see Section 6.2); Note: If necessary, the incidental use of non-steroidal anti-inflammatory drugs (NSAIDs) and paracetamol (2 g/day, 10 g/week) may be acceptable at the Investigator's discretion and will be documented in the eSource system. The use of nutritional supplements during this time that are not believed to have the potential to affect participant safety nor the overall results of the study, may be permitted on a case-by-case basis by the Investigator.

  14. Any surgical or medical condition possibly affecting drug absorption (e.g., cholecystectomy, gastrectomy, bowel disease), distribution, metabolism or excretion; 15. Personnel (e.g., Investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study; 16. Any condition that in the opinion of the Investigator would jeopardise the safety or rights of a person participating in the study or would render the person unable to comply with the protocol; 17. Personal history of malaria; 18. Volunteer has travelled to or lived in a malaria-endemic area within 6 months prior to planned study enrolment; 19. Plans to travel to malaria-endemic region during the study period up to last follow-up visit; 20. Previous participation in any malaria vaccine or Controlled Human Malaria Infection (CHMI) study/VIS; 21. Falling in moderate or higher risk category for a fatal or non-fatal cardiovascular event within 5 years (> 5%) determined by a validated risk estimation system, e.g., SCORE [21]; 22. Use of systemic antibiotics with known antimalarial activity within 5 half-lives of PfSPZ-DVI Challenge (e.g., trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones or azithromycin) or an anticipated requirement for the use of these during the study period (see Section 6.2); 23. Receipt of blood or blood-derived products (including immunoglobulin) within 3 months prior to screening. Receipt of packed RBCs given for an emergent indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed RBCs emergently given during an elective surgery).

Note: In case of an out-of-range clinical laboratory test (according to the clinically acceptable ranges for study inclusion laboratory tests in Attachment 4), vital sign or ECG value that will determine a participant's eligibility, or in case of a positive drug screen, a retest or expert evaluation can be requested. Results of any retest must be available prior to inoculation. The result of the retest will be considered for participant eligibility at the Investigator's discretion. Participants can be rescreened at the discretion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Chughlay, MD, Study Director — Medicines for Malaria Venture
Locations (1):
- SGS Belgium NV Clinical Pharmacology Unit, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1: 8 healthy, malaria-naïve males and females, aged 18-55 years, will be enrolled. The target level of parasitaemia, previously achieved in healthy participants enrolled in malaria VIS at other study sites (see Section 3.2), is 5000 parasites/mL blood in Cohort 1.
  qPCR will be performed and malaria clinical score assessed twice daily and participants will be administered registered antimalarial therapy, i.e., Riamet® (see Section 5.1), when the following criteria are met: Cohort 1: ≥5000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
  Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet: artemether-lumefantrine 6 x of 4 tablets at approximately 0, 8, 24, 36, 48 and 60 h
  PfSPZ-DVI Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
- PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2: 8 healthy, malaria-naïve males and females, aged 18-55 years, will be enrolled. The target level of parasitaemia, previously achieved in healthy participants enrolled in malaria VIS at other study sites (see Section 3.2), is 10000 parasites/mL blood in Cohort 2.
  qPCR will be performed and malaria clinical score assessed twice daily and participants will be administered registered antimalarial therapy, i.e., Riamet® (see Section 5.1), when the following criteria are met: Cohort 2: ≥10000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
  Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet: artemether-lumefantrine 6 x of 4 tablets at approximately 0, 8, 24, 36, 48 and 60 h
  PfSPZ-DVI Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
Period: Overall Study
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1: 8 healthy, malaria-naïve males and females, aged 18-55 years, will be enrolled per cohort; a participant may be enrolled in one cohort only. The target level of parasitaemia for cohort 1, previously achieved in healthy participants enrolled in malaria VIS at other study sites, is 5000 parasites/mL blood.
  qPCR will be performed and malaria clinical score assessed twice daily and participants will be administered registered antimalarial therapy, i.e., Riamet®, when the following criteria are met:
  Cohort 1: ≥5000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
  Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet: artemether-lumefantrine 6 x of 4 tablets at approximately 0, 8, 24, 36, 48 and 60 h
  PfSPZ-DVI Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
- PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2: 8 healthy, malaria-naïve males and females, aged 18-55 years, will be enrolled per cohort; a participant may be enrolled in one cohort only. The target level of parasitaemia for cohort 2, previously achieved in healthy participants enrolled in malaria VIS at other study sites, is 10,000 parasites/mL blood.
  qPCR will be performed and malaria clinical score assessed twice daily and participants will be administered registered antimalarial therapy, i.e., Riamet®, when the following criteria are met:
  Cohort 2: ≥10000 parasites/mL blood or earlier if a participant has a malaria clinical score >6 or at Investigator's discretion.
  Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet: artemether-lumefantrine 6 x of 4 tablets at approximately 0, 8, 24, 36, 48 and 60 h
  PfSPZ-DVI Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
- Total: Total of all reporting groups
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (9.3) | 43.1 (9.2) | 42.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Observed or Self-reported Adverse Events (AEs) Considered PfSPZ-DVI Challenge Inoculum-related.
Description: Based on their start date(time), AEs will be allocated to the phase during which they started (Screening, Challenge, Rescue). Each AE will therefore be reported in only one phase.
Time Frame: Screening until end of study, day 28.
Measure: Number; unit: Incidence
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
Incidence
  Adverse events | 13 | 12
  Any grade 3 or more adverse event | 1 | 2
  Screening Adverse events | 0 | 0
  Challenge adverse events | 7 | 5
  Challenge adverse events grade 3 or above | 0 | 0
  Rescue adverse events | 6 | 7
  Rescue adverse events grade 3 or above | 1 | 2

2. Primary Outcome: Change in Malaria Clinical Score From PfSPZ-DVI Challenge Until Parasite Clearance.
Description: Malaria Clinical Score
  14 signs/symptoms frequently associated with malaria will be graded using a 4-point scale (absent: 0; mild: 1; moderate: 2; severe: 3): headache, myalgia (muscle ache), arthralgia (joint ache), fatigue/lethargy, malaise (general discomfort/uneasiness), chills/shivering/rigors, sweating/hot spells, anorexia, nausea, vomiting, abdominal discomfort, fever, tachycardia and hypotension.
  Malaria clinical score is calculated as the sum of all (14) malaria sign and symptoms scores (maximum score is 42).
Time Frame: Day 1 until end of study, day 28.
Population: Safety set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
score on a scale | 9.63 (7.82) | 13.0 (1.69)

3. Primary Outcome: Time to First PCR Positivity.
Description: For the purpose of this study, 'PCR positivity' is used for the 'protocol-defined PCR positivity'
Time Frame: Day 1 to day 21
Population: PD analysis set: subjects from the safety analysis set with at least one available PD data who received all Riamet® doses and who experienced no major protocol deviations with relevant impact on PD data
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
Days | 9.76 [8.58 to 11.11] | 9.60 [8.86 to 10.41]

4. Primary Outcome: Parasitaemia at First PCR Positivity
Description: POSITIVE PARASITAEMIA IS DEFINED AS qPCR OUTCOME >=250 PARASITES per mL BLOOD.
Time Frame: Day 1 to day 21
Population: ANALYSIS set: PD
Measure: Geometric Mean (95% Confidence Interval); unit: PARASITES/mL
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
PARASITES/mL | 367.2 [280.0 to 481.5] | 711.7 [405.7 to 1248.5]

5. Primary Outcome: Time to Parasitaemia of ≥5000 Parasites Per mL Blood (Cohorts 1 and 2)
Time Frame: Day 1 to day 21
Population: ANALYSIS SET: PD
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
Days | 11.19 [10.42 to 12.42] | 11.46 [10.96 to 12.42]

6. Primary Outcome: Parasitaemia at the Time Parasitaemia ≥5000 Parasites Per mL Blood (Cohorts 1 and 2)
Time Frame: Day 1 to day 21
Population: ANALYSIS SET: PD
Measure: Geometric Mean (95% Confidence Interval); unit: PARASITES/mL
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
PARASITES/mL | 12807.4 [7736.0 to 21203.4] | 18831.7 [8739.3 to 40578.9]

7. Primary Outcome: Time to First Dose of Treatment With Artemether-lumefantrine (Riamet®) (Cohorts 1 and 2)
Time Frame: Day 1 to day 21
Population: ANALYSIS SET: PD
Measure: Geometric Mean (95% Confidence Interval); unit: Days
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
Days | 12.09 [10.97 to 13.32] | 12.04 [11.46 to 12.65]

8. Primary Outcome: Parasitaemia at First Dose of Treatment With Riamet® (Cohorts 1 and 2)
Time Frame: Day 1 to day 21
Population: ANALYSIS SET: PD
Measure: Geometric Mean (95% Confidence Interval); unit: PARASITES/mL
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
PARASITES/mL | 3936.7 [218.6 to 70890.4] | 9454.3 [3662.0 to 24408.5]

9. Primary Outcome: Incidence of Positive PCR and Parasitaemia of ≥5000 Parasites Per mL Blood.
Time Frame: Day 1 with PfSPZ-DVI Challenge and Day 28 (per cohort).
Population: ANALYSIS SET: PD
Measure: Count of Participants; unit: Participants
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
Number analyzed (Participants) | 8 | 8
Participants | 8 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously from informed consent at the Screening visit (Day -28 to Day -2) until the last study-related activity at the End Of Study Visit (Day 28).
Description: At regular intervals during the study, participants were asked non-leading questions to determine the occurrence of any AEs. All AEs reported spontaneously during the course of the study were recorded as well.
Arm/Group | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 1 (N=8) | PfSPZ-DVI Challenge and Artemether Lumefantrine Cohort 2 (N=8)
Influenza like illness (Flu-like Symptoms) (General disorders) | 7 (10) | 8 (8)
Injection site warmth (General disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This exploratory study focused on the methodology of malaria inoculation in healthy participants. No formal sample size calculation was performed.

No formal statistical analysis was performed for the primary endpoint "Changes from baseline in haematology, clinical chemistry and urinalysis parameters, vital signs and electrocardiogram (ECG) parameters". A qualitative interpretation is available if requested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No announcement, oral presentation or publication relating to the Services shall be made by SGS without the prior written approval of Sponsor, except as may be otherwise required by law.

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT04310085/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT04310085/SAP_001.pdf